CLINICAL TRIAL: NCT03434119
Title: A 26-week Randomized, Open-label, Active-controlled, 2-treatment Arm, Parallel Group Multi-center Study, Comparing the Efficacy and Safety of Soliqua™100/33 Versus Lantus® in Ethnically/Racially Diverse Patients With Type 2 Diabetes Mellitus Inadequately Controlled on Basal Insulin and Oral Antidiabetic Agents
Brief Title: Efficacy and Safety of Soliqua Versus Lantus in Ethnically/Racially Diverse Patients With Type 2 Diabetes Mellitus Inadequately Controlled on Basal Insulin and Oral Antidiabetic Agents
Acronym: LixiLan-D
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: ("Trial terminated (recruitment delays)")
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LPS14860; U1111-1200-1891 (Other: UTN)
Record Dates: First submitted 2018-02-09; First posted 2018-02-15 (Actual); Results first posted 2020-01-13 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine; lixisenatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Soliqua 100/33 (Experimental): Soliqua 100/33 (Insulin glargine/lixisenatide) once daily in the morning within 1 hour before breakfast, on top of oral anti-diabetic drug (OAD) therapy for 26 weeks.
  Interventions: Drug: Insulin glargine/Lixisenatide; Drug: Background therapy
- Lantus (Active Comparator): Lantus (Insulin glargine) once daily at any time of the day but at about the same time every day on top of OAD therapy for 26 weeks.
  Interventions: Drug: Insulin glargine (HOE901); Drug: Background therapy

INTERVENTIONS:
Drug: Insulin glargine/Lixisenatide — Insulin glargine (100 units per milliliter [U/mL]) and lixisenatide (33 micrograms per milliliter [mcg/mL]) self administered by a subcutaneous injection using a prefilled pen. Dose was individually titrated to achieve target fasting self-monitoring of plasma glucose (SMPG) of 80 to 100 milligrams per deciliter (mg/dL) (4.4 to 5.6 millimoles per liter [mmol/L]) while avoiding hypoglycemia.
  Other Names: Soliqua 100/33; HOE901/AVE0010
  Arms: Soliqua 100/33
Drug: Insulin glargine (HOE901) — Insulin glargine 100 U/mL self-administered by a subcutaneous injection using a prefilled pen. Dose was individually titrated to achieve target fasting SMPG of 80 to 100 mg/dL (4.4 to 5.6 mmol/L) while avoiding hypoglycemia.
  Other Names: Lantus; HOE901
  Arms: Lantus
Drug: Background therapy — Oral Anti diabetics Drugs (OADs) administered orally according to the locally approved label.

SUMMARY:
Primary Objective:

* To demonstrate the superiority of Soliqua 100/33 versus Lantus in the hemoglobin A1c (HbA1c) change within the overall population.
* To demonstrate the benefit of Soliqua 100/33 versus Lantus in the HbA1c within each ethnic/racial subgroup evaluated (ie, Hispanics of any race, non-Hispanic black/African Americans and non-Hispanic Asians).

Secondary Objective:

* To assess the effects of Soliqua 100/33 versus Lantus on the secondary efficacy parameters within each ethnic/racial subgroup evaluated.
* To assess the change in daily insulin glargine dose within each ethnic/racial subgroup.
* To evaluate the safety and tolerability (e.g., gastrointestinal tolerability) of Soliqua 100/33 versus Lantus within each ethnic/racial subgroup.

DETAILED DESCRIPTION:
The study duration was approximately 29 weeks including 2 weeks screening period, 26 weeks open label treatment period, and a 3 days follow-up period.

ELIGIBILITY:
Inclusion criteria :

* Participants with type 2 diabetes mellitus (T2DM) diagnosed at least 1 year prior to the screening visit (signing of informed consent).
* Uncontrolled diabetes as demonstrated by a screening centrally measured hemoglobin A1c (HbA1c) between 7.5% and 10% (inclusive).
* Participants who were Hispanics of any race, non-Hispanic black/African Americans or non-Hispanic Asians. Note: Decision for ethnic/racial inclusion was made based on the participant's self-identification. Mixed-race participants must select 1 of the above-mentioned categories. If such selection could not be made, the candidate would be ineligible to participate in the study.
* Participants who had been treated with any basal insulin (ie, glargine - U100 or U300, detemir, degludec, intermediate-acting [human Neutral Protamine Hagedorn (NPH]) for at least 6 months prior to Visit 1.
* The basal insulin regimen (ie, type of insulin and time/frequency of the injection) had been stable for at least 3 months prior to Visit 1.
* The basal insulin dose had been stable (defined as up to ±20% [1/5 of the dose] variability) for at least 2 months prior to Visit 1 within the following dose ranges:
* 15 to 50 units/day if HbA1c at Visit 1 is less than or equal to (<=)8.5%, and
* 15 to 40 units/day if HbA1c at Visit 1 is greater than (>)8.5%.
* Participants receiving 1 or 2 of the following OAD drugs: metformin, pioglitazone/rosiglitazone, an sodium-glucose transport protein 2 (SGLT-2) inhibitor or a sulfonylurea (SU), at stable doses for at least 12 weeks prior to Visit 1.

Exclusion criteria:

* Age <18 years of age at Visit 1.
* A body mass index (BMI) <=20 or >40 kg/m^2 at Visit 1.
* Fasting plasma glucose (FPG) >200 mg/dL (by central lab measurement) at Visit 1 (1-time repeat measurement before Visit 2 is permitted).
* Type 1 DM or any diabetes other than T2DM.
* Any use of OAD drugs other than those described in the inclusion criteria (e.g., but not limited to, glucagon like peptide-1 receptor agonist (GLP-1 RA), dipeptidyl peptidase 4 (DPP4) inhibitors) within 12 weeks prior Visit 1.
* Use of any other type of insulin except for basal insulin (e.g., prandial or premixed insulin, insulin pump) within 6 months prior to Visit 1. Note: History of short-term treatment (i.e, <=10 days) with other insulin types due to intercurrent illness was permitted at the discretion of the Investigator.
* Known history of discontinuation of treatment with a GLP-1 RA due to safety/tolerability reasons.
* Use of systemic glucocorticoids for a total duration of >7 days within 12 weeks prior to Visit 1.
* Initiation/change in type or dose of a weight loss drug within 12 weeks prior to Visit 1.

The above information is not intended to contain all considerations relevant to a participants's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 241 (Actual)
Dates: Start 2018-02-20 (Actual); Primary Completion 2019-01-07 (Actual); Study Completion 2019-01-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (85):
- United States (85):
  - Investigational Site Number 8400072, Montgomery, Alabama
  - Investigational Site Number 8400077, Little Rock, Arkansas
  - Investigational Site Number 8400095, Little Rock, Arkansas
  - Investigational Site Number 8400013, Little Rock, Arkansas
  - Investigational Site Number 8400076, Anaheim, California
  - Investigational Site Number 8400052, Anaheim, California
  - Investigational Site Number 8400069, Anaheim, California
  - Investigational Site Number 8400060, Burbank, California
  - Investigational Site Number 8400049, Cerritos, California
  - Investigational Site Number 8400078, Chula Vista, California
  - Investigational Site Number 8400047, Escondido, California
  - Investigational Site Number 8400066, Fountain Valley, California
  - Investigational Site Number 8400050, Greenbrae, California
  - Investigational Site Number 8400092, Huntington Park, California
  - Investigational Site Number 8400015, Los Angeles, California
  - Investigational Site Number 8400011, Los Angeles, California
  - Investigational Site Number 8400301, Los Angeles, California
  - Investigational Site Number 8400302, Los Angeles, California
  - Investigational Site Number 8400303, Los Angeles, California
  - Investigational Site Number 8400304, Los Angeles, California
  - Investigational Site Number 8400006, Los Gatos, California
  - Investigational Site Number 8400048, Oakland, California
  - Investigational Site Number 8400053, Orange, California
  - Investigational Site Number 8400084, Pomona, California
  - Investigational Site Number 8400081, Pomona, California
  - Investigational Site Number 8400042, Rancho Cucamonga, California
  - Investigational Site Number 8400063, San Carlos, California
  - Investigational Site Number 8400091, San Diego, California
  - Investigational Site Number 8400086, San Jose, California
  - Investigational Site Number 8400074, Santa Ana, California
  - Investigational Site Number 8400037, Temecula, California
  - Investigational Site Number 8400087, Vallejo, California
  - Investigational Site Number 8400024, Van Nuys, California
  - Investigational Site Number 8400007, Ventura, California
  - Investigational Site Number 8400054, Englewood, Colorado
  - Investigational Site Number 8400023, Hamden, Connecticut
  - Investigational Site Number 8400041, Gainesville, Florida
  - Investigational Site Number 8400075, Jacksonville, Florida
  - Investigational Site Number 8400036, Miami, Florida
  - Investigational Site Number 8400017, Miami, Florida
  - Investigational Site Number 8400016, Miami Lakes, Florida
  - Investigational Site Number 8400014, Ocoee, Florida
  - Investigational Site Number 8400028, Port Charlotte, Florida
  - Investigational Site Number 8400097, St. Petersburg, Florida
  - Investigational Site Number 8400035, St. Petersburg, Florida
  - Investigational Site Number 8400094, Tampa, Florida
  - Investigational Site Number 8400025, Atlanta, Georgia
  - Investigational Site Number 8400051, Atlanta, Georgia
  - Investigational Site Number 8400093, Atlanta, Georgia
  - Investigational Site Number 8400005, Savannah, Georgia
  - Investigational Site Number 8400038, Chicago, Illinois
  - Investigational Site Number 8400088, Chicago, Illinois
  - Investigational Site Number 8400031, Des Plaines, Illinois
  - Investigational Site Number 8400064, Evanston, Illinois
  - Investigational Site Number 8400057, Gurnee, Illinois
  - Investigational Site Number 8400030, Gretna, Louisiana
  - Investigational Site Number 8400009, New Orleans, Louisiana
  - Investigational Site Number 8400065, Baltimore, Maryland
  - Investigational Site Number 8400061, Rockville, Maryland
  - Investigational Site Number 8400079, Chelsea, Michigan
  - Investigational Site Number 8400001, Flint, Michigan
  - Investigational Site Number 8400012, Flint, Michigan
  - Investigational Site Number 8400090, Las Vegas, Nevada
  - Investigational Site Number 8400082, Las Vegas, Nevada
  - Investigational Site Number 8400018, Linden, New Jersey
  - Investigational Site Number 8400003, The Bronx, New York
  - Investigational Site Number 8400062, Philadelphia, Pennsylvania
  - Investigational Site Number 8400043, Columbia, South Carolina
  - Investigational Site Number 8400021, Dallas, Texas
  - Investigational Site Number 8400040, Fort Worth, Texas
  - Investigational Site Number 8400045, Houston, Texas
  - Investigational Site Number 8400002, Humble, Texas
  - Investigational Site Number 8400039, Kerrville, Texas
  - Investigational Site Number 8400096, Lufkin, Texas
  - Investigational Site Number 8400027, San Antonio, Texas
  - Investigational Site Number 8400083, San Antonio, Texas
  - Investigational Site Number 8400008, Splendora, Texas
  - Investigational Site Number 8400055, Spring, Texas
  - Investigational Site Number 8400070, Sugar Land, Texas
  - Investigational Site Number 8400085, Sugar Land, Texas
  - Investigational Site Number 8400059, Webster, Texas
  - Investigational Site Number 8400044, Manassas, Virginia
  - Investigational Site Number 8400068, Norfolk, Virginia
  - Investigational Site Number 8400033, Richmond, Virginia
  - Investigational Site Number 8400029, Richland, Washington

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 94 sites in United States (US). A total of 534 participants were screened between 20 February 2018 and 01 November 2018, of which 293 participants were screen failures. Screen failures were mainly due to glycated hemoglobin A1c (HbA1c) level less than (<)7.5% or greater than (>)10% at the screening visit.
Pre-assignment Details: Randomization was stratified by self-reported ethnic/racial group, screening HbA1c values (<8.5% vs >=8.5%), background use of sodium-glucose co-transporter-2 (SGLT-2) inhibitors (yes/no), background use of sulfonylureas (yes/no). Assignment to arms was done centrally by an interactive response technology (IRT) in 1:1 ratio (Soliqua 100/33:Lantus).
Period: Overall Study
Arm/Group | Soliqua 100/33 | Lantus
Started | 116 | 125
Treated | 115 | 125
Completed | 9 | 12
Not Completed | 107 | 113
Not completed — Randomized but not treated | 1 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Poor Compliance to Protocol | 0 | 1
Not completed — Study Terminated by Sponsor | 91 | 102
Not completed — Withdrawal by Subject | 7 | 5
Not completed — Other than specified | 7 | 5

BASELINE CHARACTERISTICS:
Population: Analysis was performed on randomized population.
Groups:
- Soliqua 100/33: Soliqua 100/33 (Insulin glargine/lixisenatide) once daily in the morning within 1 hour before breakfast, on top of OAD therapy for 26 weeks.
- Total: Total of all reporting groups
Arm/Group | Soliqua 100/33 | Lantus | Total
Number analyzed (Participants) | 116 | 125 | 241
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.6 (9.7) | 57.7 (11.9) | 59.6 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 67 | 124
  Male | 59 | 58 | 117
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanics of any race | 60 | 64 | 124
  Non-Hispanic black or African Americans | 39 | 40 | 79
  Non-Hispanic Asians | 17 | 21 | 38
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] | 30.90 (4.74) | 30.67 (4.93) | 30.78 (4.83)
Duration of Diabetes [Count of Participants; unit: Participants]
  <10 years | 26 | 39 | 65
  >=10 years | 90 | 86 | 176
Glycated Haemoglobin (HbA1c %) [Mean (Standard Deviation); unit: percentage of hemoglobin] — Population: Number of participants analyzed = participants with available data for specified measure.
  percentage of hemoglobin
    number analyzed (Participants) | 114 | 125 | 239
    (all) | 8.62 (0.74) | 8.62 (0.68) | 8.62 (0.71)
Body Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 84.97 (15.89) | 84.84 (19.34) | 84.90 (17.73)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Glycated Hemoglobin (HbA1c) at Week 26
Description: Change in HbA1c was calculated by subtracting baseline value from Week 26 value.
Time Frame: Baseline, Week 26
Population: Analysis was performed on intent-to-treat (ITT) population that included all randomized participants. Here, overall number of participants analyzed = participants with available data for the specified outcome measure.
Measure: Mean (Standard Deviation); unit: percentage of HbA1c
Arm/Group | Soliqua 100/33 | Lantus
Number analyzed (Participants) | 19 | 26
percentage of HbA1c | -1.86 (0.96) | -1.07 (1.17)

2. Secondary Outcome: Percentage of Participants Achieving HbA1c Target of <7% at Week 26
Description: Participants who had no available assessment for HbA1c at Week 26 were considered as non-responders.
Time Frame: Week 26
Population: Analysis was performed on ITT population. Here, overall number of participants analyzed = participants with available data for the specified outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Soliqua 100/33 | Lantus
Number analyzed (Participants) | 19 | 26
percentage of participants | 52.6 | 30.8

3. Secondary Outcome: Change From Baseline in 2-hour Postprandial Glucose (PPG) Following a Standardized Mixed Meal at Week 26
Description: The 2-hour PPG test measured blood glucose 2 hours after eating a standardized breakfast meal.
Time Frame: Baseline, Week 26
Population: Data were not collected, hence planned analysis was not performed due to early termination of the study.
Arm/Group | Soliqua 100/33 | Lantus
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Change From Baseline in 2-Hour Blood Glucose Excursion During Standardized Meal Test at Week 26
Time Frame: Baseline, Week 26
Population: Data were not collected, hence planned analysis was not performed due to early termination of the study.
Arm/Group | Soliqua 100/33 | Lantus
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change From Baseline in Daily Insulin Glargine Dose at Week 26
Description: Change in daily dose was calculated by subtracting baseline value from Week 26 value.
Time Frame: Baseline, Week 26
Population: Analysis was performed on ITT population. Here, overall number of participants analyzed = participants with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: International Units (IU)
Arm/Group | Soliqua 100/33 | Lantus
Number analyzed (Participants) | 9 | 11
International Units (IU) | 18.7 (16.4) | 14.1 (16.5)

6. Secondary Outcome: Change From Baseline in Body Weight at Week 26
Description: Change in body weight was calculated by subtracting baseline value from Week 26 value.
Time Frame: Baseline, Week 26
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: kilograms (kg)
Arm/Group | Soliqua 100/33 | Lantus
Number analyzed (Participants) | 18 | 24
kilograms (kg) | 1.69 (3.74) | 1.52 (2.92)

7. Secondary Outcome: Percentage of Participants With Hypoglycemic Events (Any Hypoglycemia, Severe Hypoglycemia, Documented Hypoglycemia) During the On-Treatment Period
Description: Severe hypoglycemia was an event in which the participant required the assistance of another person to actively administer carbohydrate, glucagon, or other resuscitative actions. Documented hypoglycemia with plasma glucose cut-off of <=70 mg/dL (3.9 mmol/L) was any hypoglycemia documented by a measured plasma glucose <=70 mg/dL (3.9 mmol/L) and excluding plasma glucose <54 mg/dL regardless of symptoms. Documented hypoglycemia with plasma glucose cut-off of <54 mg/dL (3.0 mmol/L) was any hypoglycemia documented by a measured plasma glucose <54 mg/dL (3.0 mmol/L) regardless of symptoms.
Time Frame: Baseline to Week 26
Population: Analysis was performed on safety population that included all randomized participants who received at least 1 dose of open-label investigational medicinal product (IMP), regardless of the amount of treatment administered. Participants were analyzed according to the treatment actually received.
Measure: Number; unit: percentage of participants
Arm/Group | Soliqua 100/33 | Lantus
Number analyzed (Participants) | 115 | 125
percentage of participants
  Any hypoglycemia | 48.7 | 52.8
  Severe hypoglycemia | 1.7 | 2.4
  Documented hypoglycaemia <=70 mg/dL (3.9 mmol/L) | 43.5 | 48.8
  Documented hypoglycaemia <54 mg/dL (3.0 mmol/L) | 12.2 | 18.4

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs) were collected from signature of the informed consent form up to the final visit (maximum treatment exposure: 194 days) regardless of seriousness or relationship to investigational product.
Description: Reported AEs and deaths are treatment emergent AEs that is AEs that developed/worsened or became serious and deaths that occurred during the 'on treatment period' (the time from the first injection of IMP up to 3 days after the last injection of IMP, regardless of the introduction of rescue therapy). Analysis was performed on safety population.
Arm/Group | Soliqua 100/33 | Lantus
All-Cause Mortality (participants affected / at risk) | 0/115 | 0/125
Serious Adverse Events (participants affected / at risk) | 7/115 | 4/125
Other Adverse Events (participants affected / at risk) | 21/115 | 20/125
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Soliqua 100/33 (N=115) | Lantus (N=125)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute Myocardial Infarction (Cardiac disorders) | 1 (1) | 0 (0)
Angina Unstable (Cardiac disorders) | 0 (0) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac Failure Congestive (Cardiac disorders) | 1 (1) | 0 (0)
Coronary Artery Disease (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial Infarction (Cardiac disorders) | 1 (1) | 0 (0)
Rectal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastroenteritis Viral (Infections and infestations) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Invasive Ductal Breast Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Facial Paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Hypoglycaemic Unconsciousness (Nervous system disorders) | 0 (0) | 1 (1)
Alcohol Withdrawal Syndrome (Psychiatric disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Soliqua 100/33 (N=115) | Lantus (N=125)
Diarrhoea (Gastrointestinal disorders) | 8 (13) | 3 (4)
Nausea (Gastrointestinal disorders) | 8 (12) | 2 (2)
Vomiting (Gastrointestinal disorders) | 6 (7) | 2 (2)
Upper Respiratory Tract Infection (Infections and infestations) | 3 (3) | 10 (11)
Headache (Nervous system disorders) | 7 (11) | 8 (12)

LIMITATIONS AND CAVEATS:
Planned analysis could not be performed due to early study termination.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2017-12-18): https://cdn.clinicaltrials.gov/large-docs/19/NCT03434119/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-28): https://cdn.clinicaltrials.gov/large-docs/19/NCT03434119/SAP_001.pdf